CLINICAL TRIAL: NCT04166253
Title: The Potential Protective Effects of Vitamin (D) Against Doxorubicin Induced Cardiotoxicity in Breast Cancer Patients
Brief Title: Protective Role of Vitamin D in Breast Cancer Patients Treated With Doxorubicin
Acronym: VDDOXO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Noha El Bassiouny, Lecturer of clinical pharmacy, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 919PP17
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vitamin D; alfacalcidol

STUDY DESIGN:
Intervention Model Description: 2 arms one is a control arm recieving only doxorubucin adjuvant chemotherapy and another intervention arm recieving doxorubucin as well as vitamin D orally once daily for 3 months
Who Masked: Participant
Masking Description: The participant did not know the exact drug he is using.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (No Intervention): Control group of breast cancer patients will receive adjuvant AC chemotherapy
- Vitamin D group (Experimental): Intervention group of breast cancer patients will receive adjuvant AC chemotherapy in addition to vitamin D (alfacalcidol 0.5 mcg orally once daily
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Alfacalcidol oral tablets once daily
  Other Names: Alfacalcidol
  Arms: Vitamin D group

SUMMARY:
The study is aimed at Evaluation of the potential protective effect of Vitamin D in doxorubucin- induced toxicity in breast cancer patients.

Proposal Steps:

1. 100 Patients recruited from Alexandria Main University Hospital (AMUH), Oncology Unit are randomly assigned in to two groups:

   * Control group (n=50) the patient will receive AC regimen (Doxorubucin & cyclophosphamide) for 4 cycles every 21 day (i.e. 3 months.)
   * Vitamin D group (n=50) who will receive 4 Cycles AC regimen in addition to vitamin D (Bon One 0.5 microgram®) once daily.
2. Echocardiography (Echo) will be done at base line and at the end of the treatment.
3. Vitamin D, LDH, Troponin-t as well as IL-6 will be assessed at baseline and at the end of the study.

DETAILED DESCRIPTION:
Research Objectives: Evaluation of the potential protective effect of Vitamin D in doxorubucin- induced toxicity in breast cancer patients.

Proposal Steps:

1. Assessing breast cancer patients taking part in the study receiving adjuvant chemotherapy AC (Anthracycline (Doxorubucin)-cyclophosphamide) for breast cancer for 4 cycles every 21 day (i.e. 3 months.)
2. 100 Patients are randomly assigned in to two groups:

   * Control group (n=50) the patient will receive AC regimen (Doxorubucin & Cyclophosphamide) for 4 cycles every 21 day (i.e. 3 months.)
   * Vitamin D group (n=50) who will receive 4 Cycles AC regimen in addition to vitamin D once daily.
3. All participants are recruited from AMUH Hospital Oncology Unit. All participants will be given their consent. The study will be approved by research ethics committee of Damanhour University.
4. Tumor staging is done according to American joint committee on cancer (TNM staging of breast cancer eighth edition (Amin et al., 2017).
5. All patients will be submitted to:

   * Full patient history and clinical examination.
   * Routine follow up before and after each chemotherapy cycle (complete blood picture, liver function tests, renal function tests.
6. Echocardiography (Echo) at base line and at the end of the treatment.
7. Vitamin D, LDH, Troponin-t as well as IL-6 will be assessed at baseline and at the end of the study.

Methodology:

Venous blood samples will be analyzed using ELISA Vitamin D, IL-6 kits and immuno-histo-chemistry Troponoin-T and LDH and kits.

ELIGIBILITY:
Inclusion Criteria:

* Patients has a good performance status (ECOG 0-2) according to eastern cooperative oncology group (ECOG) score.
* Adequate complete blood picture patients.
* Females from (30-65) years of old.
* Normal renal and liver functions.

Exclusion criteria:

* Cardiac diseased or reduced cardiac output with left ventricular ejection fraction less than 50%.
* Hepatic impaired patients.
* Pregnancy or breast feeding or child bearing state.
* Patient with history of allergy to vitamin D.
* Concomitant use of other vitamins.
* Renal impaired patients.
* History of breast cancer.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Troponin-T in ng/l | 3 months
  A change in plasma levels of Troponin-T in ng/l
Vitamin D in ng/ml | 3 months
  A change in plasma levels of Vitamin D in ng / ml
LDH in U/L | 3 months
  A change in plasma levels of LDH in U/L
Interleukin-6 in MIU/ml | 3 months
  A change in plasma levels of Interleukin-6 in MIU/ ml

CONTACTS AND LOCATIONS:
Overall Officials: Maged W Helmy, PhD, Study Director — Professor of Pharmacology, Faculty of pharmacy, Damanhour University; Gehan A Khedr, PhD, Study Director — Assistant Professor of Oncology, Faculty of Medicine, Alexandria University; Noha A El Bassiouny, PhD, Study Director — Lecturer of Clinical Pharmacy, Faculty of Pharmacy, Damanhour University; Mostafa A Mahmoud, PharmD, Principal Investigator — Clinical Pharmacy Specialist
Locations (1):
- Damnhour university, Beheira, Egypt

IPD SHARING:
Plan to Share IPD: No
Summary of data